CLINICAL TRIAL: NCT02973477
Title: Dapagliflozin and Measures of Cardiovascular Autonomic Function in Patients With Type 2 Diabetes (T2D)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00121107
Record Dates: First submitted 2016-11-16; First posted 2016-11-25 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Type2 Diabetes; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — dapagliflozin; Drug Evaluation; glimepiride

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomization will be performed by the research Pharmacy. The study coordinator will not be blind to the randomization so that they can adequately discuss the medication with the participant. The study investigator will be blind to the randomization so as to not introduce bias in data qualification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Dapagliflozin/Glimepiride (Experimental): Participants will take open-label dapagliflozin 5 mg daily for 4 weeks and escalate the dose gradually up to dapagliflozin 10 mg daily as needed based on their glucose monitoring for a total of 12 weeks on dapagliflozin. Patients will then begin a 2 week washout period where they are not taking any study drugs. After the washout period, participants will receive open-label glimepiride 2 mg daily for 4 weeks and escalate the dose gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride.
  Interventions: Drug: Dapagliflozin; Drug: Glimepiride
- Group B: Glimepiride/Dapagliflozin (Experimental): Participants will take open-label glimepiride 2 mg daily for 4 weeks and escalate the dose gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride. Patients will then begin a 2 week washout period where they are not taking any study drugs. After the washout period, participants will receive open-label dapagliflozin 5 mg daily for 4 weeks and escalate the dose gradually up to dapagliflozin 10 mg daily as needed based on their glucose monitoring for a total of 12 weeks on dapagliflozin.
  Interventions: Drug: Dapagliflozin; Drug: Glimepiride

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin is a sodium glucose transporter-2 (SGLT-2) inhibitor, a new class of glucose lowering agent that reduces hyperglycemia in patients with T2D by reducing renal glucose reabsorption.
  Other Names: Study Drug
Drug: Glimepiride — Glimepiride is a sulfonylurea agent that reduces hyperglycemia in patients with T2D by stimulating insulin release from the pancreatic beta cells and reduction of glucose output from the liver.
  Other Names: Active Comparator

SUMMARY:
The purpose of this study is to evaluate the effect of dapagliflozin, a FDA approved diabetes medication, on measures of nervous system function of the heart in patients with type 2 diabetes. The investigators will compare the effect of dapagliflozin with an active comparator, glimepiride (a different FDA approved diabetes medication) on measures of heart rate variability and assess whether dapagliflozin has modulating effects on measures of nervous system function of the heart. This is a crossover study design where all participants will receive both study medications equally (12-week intervention periods) in a certain order.

DETAILED DESCRIPTION:
Study rationale: Empagliflozin and dapagliflozin are sodium-glucose transporter-2 (SGLT-2) inhibitors which prevent the reabsorption of glucose via proximal renal tubules, and are the most recently approved class for treating hyperglycemia in type 2 diabetes. Besides effective glucose lowering effects as documented by ~ 0.7-1.2% HbA1c reduction, these agents also promote weight loss and reduce blood pressure (BP). Furthermore, recent data from the Empagliflozin Cardiovascular Outcome Trial in type 2 diabetes (EMPA-REG OUTCOME) reported significant reduction in main cardiovascular disease (CVD) outcomes and CVD death in patients with type 2 diabetes (T2D). The exact mechanism of the beneficial effects on cardiovascular outcomes is not yet understood, although their effects on body weight, glucose control and BP reduction were suggested. However, other classes of drugs with similar effects such as GLP-1 receptor agonist, thiazolidinedione did not clearly show the beneficial effects in CVD outcomes. The interesting observation is that improvement in BP with SGLT-2 inhibitors occurred without a compensatory increase in HR and that most benefit was obtained also in patients with some evidence of heart failure.

Thus, the investigators postulated the hypothesis that SGLT-2 may also have a modulatory effect on the sympathetic/parasympathetic balance, and this may contribute to the potential benefits on cardiovascular outcomes in patients with diabetes.

Study Design: The investigators plan to test this hypothesis in a randomized, double-blind, 2-period crossover clinical trial comparing 12-weeks of glycemic intervention with dapagliflozin versus glimepiride. The investigators include an active comparator with glimepiride which have a similar glucose lowering in patients with T2D, to account for the effects of reductions in blood glucose on measures of CAN, and will evaluate whether changes in measures of CAN are different among patients who are taking glimepiride or dapagliflozin. The two crossover periods will be separated by a 2-week wash-out period.

All subjects will be allocated and randomized to each treatment sequence. Participants will receive blindly either dapagliflozin 5 mg or glimepiride 2 mg 1 tablet daily initially for 4 weeks then titrating the dose based on blood glucose levels up to 2 tablets daily for 8 more weeks (total 12 weeks) followed by 2-week washout period and then they will receive the study drugs in reverse order to the first period during second crossover period for 12 weeks.

Study population: 45 patients with T2D on background metformin monotherapy who are not meeting ADA recommended glycemic target.

Primary outcomes: changes in measures of cardiovascular autonomic neuropathy such as heart rate variability (HRV) as defined by frequency domain measures of HRV: low frequency (LF) power (ms2); high frequency (HF) power (ms2) as measured as LF:HF ratio.

Secondary outcomes: (i) changes in measures of HRV as defined by time domain measures of HRV: standard deviation of the normal RR interval (SDNN) (msec) and root mean square of the differences of successive RR intervals (rmsSD) (msec); (ii) changes in cardiovascular autonomic reflex tests (CARTs) as defined by: expiration/inspiration (E/I) ratio, Valsalva ratio, and 30:15 ratio; (iii) changes in measures of systolic and diastolic function will be assessed by using stress echocardiogram and evaluate the following measures: i) LVEF, ii) LV end diastolic volume, iii) LV end systolic volume, iv) LV mass, v) cardiac output.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes as defined on background metformin monotherapy who are not meeting ADA standard of care recommended glucose target.
2. Age ≥18 years

Exclusion Criteria:

1. History of multiple urinary tract infections
2. Patients with mycotic infections especially genital infections.
3. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status. This is listed as exclusion criteria but then it says that they just need careful monitoring. Is it an exclusion or not?
4. Severely hypotensive patients
5. History of unexplained microscopic or gross hematuria, or microscopic hematuria at visit 1, confirmed by a follow-up sample at next scheduled visit.
6. Presence of hypersensitivity to dapagliflozin or other SGLT2 inhibitors (e.g. anaphylaxis, angioedema, exfoliative skin conditions
7. Inability or refusal to comply with protocol
8. Current participation or participation in an experimental drug study in the previous three months
9. History of diabetic ketoacidosis
10. Planned cardiac surgery or angioplasty within 3 months
11. Recent history of acute CV events such as MI, stroke, PAD within 3 months prior to enrollment
12. Patients with severe renal impairment or unstable or rapidly progressing renal disease or end stage renal disease.
13. Clinical conditions that could interfere with the cardiovascular autonomic function and heart rate variability (arrhythmias)
14. Severe hepatic insufficiency and/or significant abnormal liver function (defined as aspartate aminotransferase >3× upper limit of normal (ULN) and/or alanine aminotransferase >3× ULN) or creatinine kinase >3× ULN.
15. History of cancer other than basal cell carcinoma and/or treatment for cancer within the last 5 years
16. Women of child-bearing potential who may be pregnant or lactating.
17. History of pancreas, kidney or liver transplant
18. History of drug or alcohol abuse
19. History of allergy to sulfa drugs
20. Presence of any condition that, in the opinion of the investigator would make it unlikely for the subject to complete the study
21. Congestive heart failure (CHF) defined as New York Heart Association class III and IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, M.D. Ph.D, Principal Investigator — University of Michigan Department of Internal Medicine Division of Metabolism, Endocrinology and Diabetes; Lynn P Ang, M.D, Principal Investigator — University of Michigan Department of Internal Medicine Division of Metabolism, Endocrinology and Diabetes
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ang L, Kidwell KM, Dillon B, Reiss J, Fang F, Leone V, Mizokami-Stout K, Pop-Busui R. Dapagliflozin and measures of cardiovascular autonomic function in patients with type 2 diabetes (T2D). J Diabetes Complications. 2021 Aug;35(8):107949. doi: 10.1016/j.jdiacomp.2021.107949. Epub 2021 May 15. PMID 34024686

RESULTS

PARTICIPANT FLOW:
Groups:
- First Dapagliflozin Then Glimepiride: Participants received open-label dapagliflozin 5 mg daily for 4 weeks and then the dose escalated gradually up to dapagliflozin 10 mg daily as needed based on their glucose monitoring for a total of 12 weeks on dapagliflozin. Patients then began a 2 week washout period where they did not take any study drugs. After the washout period, participants received open-label glimepiride 2 mg daily for 4 weeks and the dose escalated gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride.
- First Glimepiride Then Dapagliflozin: Participants received open-label glimepiride 2 mg daily for 4 weeks and the dose escalated gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride. Patients then began a 2 week washout period where they did not take any study drugs. After the washout period, participants took open-label dapagliflozin 5 mg daily for 4 weeks and then the dose escalated gradually up to dapagliflozin 10 mg daily as needed based on their glucose monitoring for a total of 12 weeks on dapagliflozin.
Period: First Intervention
Arm/Group | First Dapagliflozin Then Glimepiride | First Glimepiride Then Dapagliflozin
Started | 19 | 26
Completed | 19 | 24
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Period: Washout
Arm/Group | First Dapagliflozin Then Glimepiride | First Glimepiride Then Dapagliflozin
Started | 19 | 24
Completed | 18 | 24
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | First Dapagliflozin Then Glimepiride | First Glimepiride Then Dapagliflozin
Started | 18 | 24
Completed | 17 | 24
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First Dapagliflozin Then Glimepiride | First Glimepiride Then Dapagliflozin | Total
Number analyzed (Participants) | 19 | 26 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9) | 56 (8) | 57 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 12 | 14 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 12 | 18 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
LF:HF Ratio [Mean (Standard Deviation); unit: Ratio] — The frequency domain measures [ low-frequency (LF) power (0.04-0.15 Hz), high-frequency (HF) power (0.15-0.4 Hz), and LF:HF ratio] are obtained by spectral analysis of R-R interval from continuous electrocardiogram recordings to evaluate for sympathetic/parasympathetic (autonomic nervous function) balance. Population: 3 participants lost to follow up after baseline data collection.
  Ratio
    Baseline before First Intervention | 1.00 (1.74) | 0.73 (1.31) | 0.84 (1.49)
    Baseline before Second Intervention: number analyzed (Participants) | 18 | 24 | 42
    Baseline before Second Intervention | 0.82 (1.32) | 0.35 (1.36) | 0.61 (1.46)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Measure of Heart Rate Variability Using Dapagliflozin vs Active Comparator Glimepiride.
Description: Heart Rate Variability, as shown by the difference of the LF:HF ratio from baseline to 12 weeks per arm (two 12-week periods with a 2-week washout period. The frequency domain measures [ low-frequency (LF) power (0.04-0.15 Hz), high-frequency (HF) power (0.15-0.4 Hz), and LF:HF ratio] are obtained by spectral analysis of R-R interval from continuous electrocardiogram recordings to evaluate for sympathetic/parasympathetic (autonomic nervous function) balance.
Time Frame: from first baseline to end of 12 weeks' treatment and from second baseline (following 2 weeks of washout) to end of 12 weeks' treatment
Population: All participants who completed both interventions were included in the analysis.
Measure: Mean (Standard Deviation); unit: LF:HF ratio
Groups:
- First Dapagliflozin Then Glimepiride: Participants took open-label dapagliflozin 5 mg daily for 4 weeks and then the dose escalated gradually up to dapagliflozin 10 mg daily as needed based on their glucose monitoring for a total of 12 weeks on dapagliflozin. Patients then began a 2 week washout period where they did not take any study drugs. After the washout period, participants received open-label glimepiride 2 mg daily for 4 weeks and the dose escalated gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride.
Arm/Group | First Dapagliflozin Then Glimepiride | First Glimepiride Then Dapagliflozin
Number analyzed (Participants) | 17 | 24
LF:HF ratio
  value at 12 weeks minus value at 1st baseline | -0.18 (1.51) | -0.34 (1.54)
  value at 26 weeks minus value at 2nd baseline | 0.26 (1.85) | 0.26 (1.92)
Statistical Analysis 1: Comparison: First Dapagliflozin Then Glimepiride vs First Glimepiride Then Dapagliflozin; This is the adjusted mixed models analysis for both periods, both arms, comparing each treatment's change; Test type: Other — Mixed effects model; p = 0.28, Mixed Models Analysis — Adjusted analysis used a linear mixed effects model with unstructured covariance matrix controlled for possible period and sequence (carryover) effects for the outcome; Coefficient = 0.28, 95% CI 2-sided [-0.24 to 0.8] — The outcome was logged in the model. The outcome was the natural log of that variable and the coefficient and CI are for the relationship with the log of the outcome

2. Secondary Outcome: Changes in Measures of Heart Rate Variability (HRV) Using Dapagliflozin vs Active Comparator Glimepiride.
Description: Changes in measures of HRV as defined by: Time domain measures of HRV (continuous variables): (i) standard deviation of the normal RR interval (SDNN) (msec) and (ii) root mean square of the differences of successive RR intervals (rmsSD) (msec).
  Time domain (SDNN and rmsSD) measures of the normal R-R intervals are derived from HRV studies using a physiologic monitor (Nightingale PPM2; Zoe Medical Inc.) under paced breathing, reflecting parasympathetic activity.
  Time domain measures of the normal R-R intervals, basically reflecting parasympathetic activity, include: the difference between the longest and shortestR-R interval, standard deviation of 5-min average of normal R-R intervals (SDANN), root-mean square of the difference of successive R-R intervals (rMSSD).
Time Frame: 12 weeks on each intervention
Population: All who started an intervention were included in analysis for Before treatment. Only those who completed it are included in After treatment. Changes in numbers represent participants from an arm leaving before completing an intervention. Since 3 people who began Glimepiride did not complete it, the 44 shown in "Before" reduces to 41 "After".
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Participants Who Received Dapagliflozin Intervention: Participants received open-label dapagliflozin 5 mg daily for 4 weeks and then the dose escalated gradually up to dapagliflozin 10 mg daily as needed based on their glucose monitoring for a total of 12 weeks on dapagliflozin, whether before or after washout.
- Participants Who Received Glimepiride Intervention: Participants received open-label glimepiride 2 mg daily for 4 weeks and the dose escalated gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride whether before or after washout.
Arm/Group | Participants Who Received Dapagliflozin Intervention | Participants Who Received Glimepiride Intervention
Number analyzed (Participants) | 43 | 44
msec
  SDNN before treatment | 40.72 (16.63) | 39.75 (16.15)
  SDNN after treatment: number analyzed (Participants) | 43 | 41
  SDNN after treatment | 37.74 (16.04) | 36.46 (17.68)
  rmsSD before treatment | 26.91 (17.81) | 25.14 (13.06)
  rmsSD after treatment: number analyzed (Participants) | 43 | 41
  rmsSD after treatment | 24.30 (16.44) | 24.63 (17.38)
Statistical Analysis 1: Comparison: Participants Who Received Dapagliflozin Intervention vs Participants Who Received Glimepiride Intervention; This is the adjusted analysis to compare the difference between the values from baseline to 12 weeks between each intervention for SDNN; Test type: Other; p = 0.97, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Coefficient = -0.003, 95% CI 2-sided [-0.16 to 0.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Participants Who Received Dapagliflozin Intervention vs Participants Who Received Glimepiride Intervention; This is the adjusted analysis to compare the difference between the values from baseline to 12 weeks between each intervention for rmsSD; Test type: Other; p = 0.79, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Coefficient = -0.02, 95% CI 2-sided [-0.21 to 0.16] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Changes in Measures of Cardiac Autonomic Reflex Testing (CARTs)
Description: Changes in CARTs as defined by: i) expiration/inspiration (E/I) ratio, ii) Valsalva ratio and iii) 30:15 ratio. Cardiovascular autonomic reflex tests assess the cardiovascular autonomic function using provocative physiological maneuvers under paced breathing [R-R response to breathing (E:I ratio), to Valsalva maneuver (Valsalva ratio) and to postural changes (30:15 ratio)] at baseline and at the end of each study drug period using a physiologic monitor (Nightingale PPM2; Zoe Medical Inc.).
Time Frame: 12 weeks on each intervention
Population: All who started an intervention were included in Before rows if data was present. Only those who completed it are included in After treatment. Changes in numbers represent participants from an arm leaving before completing an intervention. Since 3 people who began Glimepiride did not complete it, the 44 shown in "Before" reduces to 41 "After".
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- All Participants Who Received Dapagliflozin: Participants received open-label dapagliflozin 5 mg daily for 4 weeks and then the dose escalated gradually up to dapagliflozin 10 mg daily as needed based on their glucose monitoring for a total of 12 weeks on dapagliflozin, whether before or after washout.
- All Participants Who Received Glimiperide: Participants received open-label glimepiride 2 mg daily for 4 weeks and the dose escalated gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride.
Arm/Group | All Participants Who Received Dapagliflozin | All Participants Who Received Glimiperide
Number analyzed (Participants) | 43 | 44
ratio
  E/I ratio before treatment | 1.13 (0.07) | 1.14 (0.08)
  EI ratio after treatment: number analyzed (Participants) | 43 | 41
  EI ratio after treatment | 1.14 (0.11) | 1.14 (0.13)
  Valsalva ratio before treatment: number analyzed (Participants) | 42 | 44
  Valsalva ratio before treatment | 1.50 (0.36) | 1.44 (0.29)
  Valsalva ratio after treatment: number analyzed (Participants) | 43 | 41
  Valsalva ratio after treatment | 1.60 (0.66) | 1.58 (0.85)
  30:15 ratio before treatment: number analyzed (Participants) | 42 | 44
  30:15 ratio before treatment | 1.17 (0.15) | 1.14 (0.09)
  30:15 ratio after treatment: number analyzed (Participants) | 43 | 41
  30:15 ratio after treatment | 1.14 (0.11) | 1.14 (0.10)
Statistical Analysis 1: Comparison: All Participants Who Received Dapagliflozin vs All Participants Who Received Glimiperide; This is the adjusted analysis for both periods, both arms, comparing each treatment's change of EI ratio; Test type: Other; p = 0.58, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Coefficient = 0.01, 95% CI 2-sided [-0.02 to 0.04]
Statistical Analysis 2: Comparison: All Participants Who Received Dapagliflozin vs All Participants Who Received Glimiperide; This is the adjusted analysis for both periods, both arms, comparing each treatment's change of Valsalva ratio; Test type: Other; p = 0.58, Mixed Models Analysis — Adjusted analysis used a linear mixed effects model with unstructured covariance matrix controlled for possible period and sequence (carryover) effects for the outcome. Coefficient provided for Valsalva ratio; Coefficient = 0.02, 95% CI 2-sided [-0.05 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: All Participants Who Received Dapagliflozin vs All Participants Who Received Glimiperide; This is the adjusted analysis for both periods, both arms, comparing each treatment's change of 30:15 ratio; Test type: Other; p = 0.56, Mixed Models Analysis — Adjusted analysis used a linear mixed effects model with unstructured covariance matrix controlled for possible period and sequence (carryover) effects for the outcome. Coefficient provided for 30:15 ratio; Coefficient = -0.01, 95% CI 2-sided [-0.05 to 0.03]

4. Secondary Outcome: Change in B-type Natriuretic Peptide With Each Intervention as a Measure of Left Ventricular Function
Description: Changes in B-type Natriuretic Peptide (BNP) with each intervention as a measure of left ventricular function.
Time Frame: 12 weeks for each intervention
Population: 1 Glimiperide-first person's BNP measurement for Before treatment was missing. Only those who completed it are included in After treatment. Changes in numbers represent participants from an arm leaving before completing an intervention. Since 2 others who began Glimepiride did not complete it, the 43 shown in "Before" reduces to 41 "After".
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- All Participants Who Received Glimepiride: Participants received open-label glimepiride 2 mg daily for 4 weeks and the dose escalated gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride.
Arm/Group | All Participants Who Received Dapagliflozin | All Participants Who Received Glimepiride
Number analyzed (Participants) | 43 | 43
pg/ml
  BNP before treatment | 12.72 (9.76) | 16.93 (13.69)
  BNP after treatment: number analyzed (Participants) | 43 | 41
  BNP after treatment | 14.76 (13.41) | 15.49 (11.58)
Statistical Analysis 1: Comparison: All Participants Who Received Dapagliflozin vs All Participants Who Received Glimepiride; This is the adjusted analysis for both periods, both arms, comparing each treatment's change of BNP; Test type: Other; p = 0.92, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Coefficient = 0.01, 95% CI 2-sided [-0.23 to 0.25]

5. Other Pre Specified Outcome: Glucose Variability
Description: Measures of glucose variability via the continuous glucose monitoring system Libre Pro
Time Frame: 2 weeks on each intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: At each study visit, patients were asked about any change in medical history or status as well as adverse events, effects, or reactions. Patients also called the study team when they experienced issues. Patients were encouraged to inform the study team if any adverse events were experienced, regardless of relatedness.
Groups:
- Dapagliflozin: Participants will take open-label dapagliflozin 5 mg daily for 4 weeks and escalate the dose gradually up to dapagliflozin 10 mg daily as needed based on their glucose monitoring for a total of 12 weeks on dapagliflozin.
- Glimepiride: Participants will take open-label glimepiride 2 mg daily for 4 weeks and escalate the dose gradually up to glimepiride 4 mg daily (no more than 4 mg daily) as needed based on their glucose monitoring for a total of 12 weeks on glimepiride.
- Not on Drug: Participants who were not on study drug, either prior to drug assignment, during washout or after ceasing taking drug prior to categorization as lost to follow up. Since all participants were definitionally present in the prior to drug assignment period, all are included here.
Arm/Group | Dapagliflozin | Glimepiride | Not on Drug
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/43 | 0/45
Other Adverse Events (participants affected / at risk) | 11/44 | 14/43 | 5/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=44) | Glimepiride (N=43) | Not on Drug (N=45)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 | 0 | 0 — Patient has a history of long airline travel
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=44) | Glimepiride (N=43) | Not on Drug (N=45)
Torn Left Hamstring (Injury, poisoning and procedural complications) | 1 | 0 | 0
Genital Yeast Infection (Infections and infestations) | 2 | 0 | 0
Cold Like Symptoms (Infections and infestations) | 2 | 0 | 1 — In Not on Drug arm, participant experienced symptoms prior to randomization
Vasovagal Episode (Nervous system disorders) | 0 | 1 | 0 — Vasovagal episode resulting in vomiting due to blood draw
Cut on Foot (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nausea, Vomiting and Dizziness (Gastrointestinal disorders) | 1 | 0 | 0
Abrasion of Left Cornea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stomach Virus (Infections and infestations) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Chest Pain (Cardiac disorders) | 0 | 1 | 0 — Nonspecific T-Wave changes on EKG - Possible relation to GERD - ED dx excluded cardiac ischemia
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — Removal of basal cell carcinoma completed
Bronchitis (Infections and infestations) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Gull Bladder Removal (Surgical and medical procedures) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Right Leg Pain and Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — Right Leg Pain and Swelling - DVT was ruled out
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Urinary Frequency and Discomfort - UTI Ruled Out (Renal and urinary disorders) | 0 | 2 | 0
Strep Throat / Tonsillitis (Infections and infestations) | 1 | 0 | 0
Diagnosis of Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Right First Metasophalangeal
Food Poisoning (Infections and infestations) | 0 | 1 | 0 — Vomiting and Diarrhea
Hypoglycemia (Endocrine disorders) | 1 | 2 | 0
Ear and Sinus Infection (Infections and infestations) | 1 | 0 | 0
Dizziness, Shakiness, Weakness and Sweaty (Endocrine disorders) | 0 | 1 | 0 — Not Hypoglycemic. Documented lowest glucose value was 92mg/dL.
Worsening Depression and Mental Fogginess (Psychiatric disorders) | 1 | 0 | 0
Pins and Needles Sensation of Lower Extremities (Nervous system disorders) | 0 | 0 | 1 — Washout post-Dapagliflozin
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Off Glimiperide due to prior Physician decision per protocol
Dizziness (Nervous system disorders) | 0 | 0 | 1 — Washout post-Glimepiride
Left Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Patient dispensed Glimepiride. Patient lost to follow up. Adverse event occurred between loss of contact and patient marked as lost to follow up
Cataract Surgery (Surgical and medical procedures) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT02973477/Prot_SAP_000.pdf